CLINICAL TRIAL: NCT05914623
Title: Effects of High-frequency Repetitive Transcranial Magnetic Stimulation on Cerebral Autoregulation in Patients With Cerebral Small Vessel Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Vice President of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMSCA-CSVD
Record Dates: First submitted 2023-06-06; First posted 2023-06-22 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Transcranial Magnetic Stimulation
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS (Active Comparator): Patients are treated with repetitive transcranial magnetic stimulation (rTMS).
  Interventions: Procedure: Repetitive transcranial magnetic stimulation
- sham-rTMS (Placebo Comparator): Patients are treated with sham repetitive transcranial magnetic stimulation (sham-rTMS).
  Interventions: Procedure: Sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Procedure: Repetitive transcranial magnetic stimulation — After enrollment, the patients received rTMS once a day for 5 consecutive days (stimulation plan: stimulation of M1 region on the affected side at 10Hz).
  Arms: rTMS
Procedure: Sham repetitive transcranial magnetic stimulation — After enrollment, the patients received sham-rTMS once a day for 5 consecutive days with the same parameters as the rTMS group, but the coil was rotated 90° away from the scalp.
  Arms: sham-rTMS

SUMMARY:
The purpose of this study was to investigate the effect of high-frequency repetitive transcranial magnetic stimulation on cerebral autoregulation in patients with cerebral small vessel disease.

DETAILED DESCRIPTION:
Current studies have shown that repetitive transcranial magnetic stimulation can change the excitability of nerve cells, improve intracerebral artery blood supply, and even reduce the degree of neurological impairment in patients with stroke. The purpose of this study was to investigate the effect of high-frequency repetitive transcranial magnetic stimulation on cerebral autoregulation in patients with cerebral small vessel disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years, regardless of gender;
2. Diagnosed with CSVD, and neuroimaging presented as recent small subcortical infarcts;
3. Initiated transcranial magnetic stimulation within 7 days of onset;
4. Subject or legal representative agreed to the treatment and signed the informed consent;

Exclusion Criteria:

1. Vascular stenosis > 50% diagnosed by Transcranial Doppler (TCD) and carotid ultrasound;
2. Previous history of atrial fibrillation or myocardial infarction within 6 months;
3. Moyamoya disease or hereditary cerebral small vessel disease, such as CADASIL;
4. White matter hyperintensities (WMH) of non-vascular origin;
5. Severe hepatic and renal diseases, cancer or other major diseases related to integral medical and surgical procedures;
6. Patients with contraindications to transcranial magnetic stimulation, such as metal or electronic devices in the brain;
7. Pregnant or breastfeeding women;
8. The patients with disorders of consciousness, agitation or insufficient bilateral temporal bone windows for insonation who cannot cooperate to dynamic cerebral autoregulation monitoring;
9. Previous history of epilepsy or family history of epilepsy;
10. Previous treatment with transcranial magnetic stimulation or its equivalent;
11. Unwillingness to be followed up or poor adherence to treatment;
12. Those who are participating in other clinical investigators, or who have participated in other clinical studies within 3 months prior to enrollment, or who have participated in this study;
13. Other conditions that the investigators deemed unsuitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-25 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
phase difference (PD) in degree | 0-5 days
  A cerebral autoregulation parameter derived from transfer function analysis. Continuous cerebral blood flow velocities of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler. Spontaneous arterial blood pressure will be simultaneously recorded using a servo-controlled plethysmograph on the left or right middle finger with an appropriate finger cuff size. Transfer function analysis will be used to derive the cerebral autoregulatory parameter.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China